CLINICAL TRIAL: NCT06385821
Title: Multicenter, Double-blind, Randomized, Parallel Group Study to Evaluate the Immunogenicity, Reactogenicity and Safety of the Grippol® Quadrivalent Vaccine in Children Aged 6 Months to 5 Years (Inclusive)
Brief Title: A Study to Prove Non-inferior Immunogenicity of Grippol Quadrivalent Compared to Grippol Plus
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NPO Petrovax (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: GriQv-ch-III-22
Record Dates: First submitted 2023-09-04; First posted 2024-04-26 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2023-11

CONDITIONS: Influenza; Influenza A; Influenza, Human; Influenza Type B; Flu; Influenza A H3N2; Influenza A H1N1; Influenza Epidemic; Flu, Human; Acute Respiratory Infection; Vaccine Reaction
Keywords: Vaccine; Influenza vaccine; acute respiratory infection
MeSH Terms: conditions — Influenza, Human; Orthomyxoviridae Infections | interventions — Grippol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Grippol Quadrivalent (Experimental): influenza quadrivalent inactivated subunit adjuvant vaccine
  Interventions: Biological: Grippol Quadrivalent
- Grippol Plus (Active Comparator): influenza trivalent inactivated polymer-subunit vaccine
  Interventions: Biological: Grippol Plus

INTERVENTIONS:
Biological: Grippol Quadrivalent — Solution for intramuscular and subcutaneous administration, 0.5 ml/dose. Children from 36 months to 5 years - in the upper third of the outer surface of the shoulder intramuscularly (in the deltoid muscle) at a dose of 0.5 ml once (Day 1). Children from 6 to 35 months - in the anterolateral surface of the thigh intramuscularly 0.25 ml twice with an interval of 3-4 weeks (Day 1, Day 25±3).
  Arms: Grippol Quadrivalent
Biological: Grippol Plus — Suspension for intramuscular and subcutaneous administration, 0.5 ml/dose. Children from 36 months to 5 years - in the upper third of the outer surface of the shoulder intramuscularly (in the deltoid muscle) at a dose of 0.5 ml once (Day 1). Children from 6 to 35 months - in the anterolateral surface of the thigh intramuscularly, 0.25 ml twice with an interval of 3-4 weeks (Day 1, Day 25±3).
  Arms: Grippol Plus

SUMMARY:
The goal of this clinical study is to prove the no less immunogenicity of the Grippol Quadrivalent vaccine compared to the Grippol plus vaccine in children aged 6 months to 5 years (inclusive) for three identical strains of the compared vaccines in terms of the "proportion of vaccinated with seroconversion in paired sera of the hemagglutination inhibition reaction obtained before and after vaccination".

DETAILED DESCRIPTION:
The main questions it aims to answer are:

1. To compare the immunogenicity of the Grippol Quadrivalent vaccine compared to the Grippol plus vaccine in children aged 6 months to 5 years (inclusive) for three identical strains of the compared vaccines in terms of "geometric mean antibody titers after vaccination"
2. Evaluate the immunogenicity of the Grippol Quadrivalent vaccine and the Grippol plus vaccine according to the following indicators:

   * Proportion of those vaccinated with seroconversion and geometric mean titer of antibodies to the fourth additional strain of compared vaccines
   * Multiplicity of the increase in the geometric mean titer of antibodies to 4 strains of the influenza virus in paired sera of the hemagglutination inhibition reaction after vaccination in relation to the initial values of antibody titers
   * Seroprotection (proportion (%) vaccinated with antibody titer ≥ 1:40 to 4 strains of influenza virus in paired sera of the hemagglutination inhibition reaction after vaccination)
3. Evaluate the effectiveness of the Grippol Quadrivalent vaccine and the Grippol plus vaccine according to the following indicators:

   * Incidence of Influenza and ARI (Month 1-Month 6 after vaccination)
   * Severity and duration of reported cases of influenza and ARI, presence of complications
4. Assess the reactogenicity of the Grippol Quadrivalent vaccine and the Grippol plus vaccine in children aged 6 months to 5 years (inclusive):

   * Frequency and nature of general and local post-vaccination reactions (7-day follow-up period after vaccine administration)
5. Assess the safety of Grippol Quadrivalent and Grippol Plus in children aged 6 months to 5 years (inclusive)

ELIGIBILITY:
Inclusion Criteria:

1. Male and female children aged 6 months to 5 years inclusive at the time of vaccination.
2. Availability of Informed consent to participate in the study, signed by one of the parents.
3. The diagnosis is "healthy", established according to standard clinical, laboratory and instrumental methods of examination carried out at screening, according to the assessment of the researcher, as well as anamnesis data (absence of acute and chronic diseases of the respiratory, cardiovascular, nervous systems, dysfunction liver or kidneys).
4. Negative result of a rapid test for SARS-CoV-2 antigen at screening.
5. For children aged 6 to 11 months inclusive: children born at gestational age ≥37 weeks weighing ≥2.5 kg.
6. Parental consent to cooperate in good faith with the investigator and center staff, attend scheduled visits, complete the self-monitoring diary, and follow the protocol.

Exclusion Criteria:

1. Vaccination with any influenza vaccine within the previous 6 months. Vaccination with other vaccines, according to the national vaccination schedule, is allowed no later than 30 days before the introduction of the study vaccine, and no earlier than 30 days after the administration of the study vaccines.
2. Participation in a clinical trial of a vaccine, medicinal product, or medical device less than 30 days prior to screening.
3. Hypersensitivity to any of the components of the studied vaccines or severe post-vaccination complications to any vaccine in history.
4. The presence at the time of screening of acute infectious diseases of any localization, or the presence of a history of acute infectious and non-infectious diseases less than 14 days before screening.
5. Body temperature in the armpit ≥37.0°C at screening or before the introduction of the vaccine.
6. History of significant chronic diseases, such as malignant neoplasms or blood diseases, autoimmune diseases, insulin-dependent diabetes mellitus, chronic diseases of the lungs, liver or kidneys, cardiovascular, nervous systems, secondary, primary and induced immunodeficiency, HIV- infections, as well as other significant, according to the researcher, diseases.
7. A history of seizures or a progressive neurological disease.
8. History of Guillain-Barré syndrome (post-infectious demyelinating polyradiculoneuropathy of autoimmune etiology).
9. Use of antipyretics, including non-steroidal anti-inflammatory drugs less than 24 hours before screening and vaccination; antibacterial drugs of systemic action - less than 72 hours before screening and vaccination; anticoagulants - less than 3 weeks before screening and vaccination; immunoglobulins, blood products - less than 3 months before screening and vaccination; long-term use of systemic corticosteroids (prednisolone or equivalent for more than 2 consecutive weeks) - less than 3 months before vaccination screening.
10. Surgery performed less than 3 months prior to screening.
11. Children of research team members or research facility staff involved in this clinical trial.
12. Orphans, children left without parental care.
13. Any other medical or social condition that, in the opinion of the investigator, precludes the participation of the child in this study.

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 824 (Actual)
Dates: Start 2022-09-21 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-10-09 (Actual)

PRIMARY OUTCOMES:
To prove non-inferior immunogenicity of the Grippol Quadrivalent vaccine when compared to the Grippol plus vaccine in children aged 6 months to 5 years (inclusive) for three matching strains of the compared vaccines | Baseline to Day 25±3
  Proportion of vaccinated seroconverters in paired hemagglutination inhibition test sera obtained before and after vaccination
  Seroconversion is defined as:
  1. increase in antibody titer to influenza virus strains to ≥ 1:40 (with initial antibody titer < 1:10); or
  2. an increase in antibody titer by 4 or more times compared to the initial titer (with an initial antibody titer ≥ 1:10) in paired sera RTGA after vaccination.
  The initial antibody titer will be the titers of antibodies to influenza virus antigens in the hemagglutination inhibition reaction obtained during screening. Post-vaccination titres will be those obtained on Day 25±3 after a single dose of vaccine in children 36 months to 5 years of age or a second dose of vaccine in children 6 to 35 months of age.

SECONDARY OUTCOMES:
Geometric mean antibody titers | Baseline to Day 25±3
  Geometric mean antibody titers after vaccination for three matching strains
Proportion of those vaccinated with seroconversion and geometric mean titer | Baseline to Day 25±3
  Proportion of those vaccinated with seroconversion and geometric mean titer of antibodies to the fourth additional strain of compared vaccines
Multiplicity of the increase in the geometric mean titer | Baseline to Day 25±3
  Multiplicity of the increase in the geometric mean titer of antibodies to 4 strains of the influenza virus in paired sera of the hemagglutination inhibition reaction after vaccination in relation to the initial values of antibody titers
Seroprotection | Baseline to Day 25±3
  Seroprotection (proportion (%) vaccinated with antibody titer ≥ 1:40 to 4 strains of influenza virus in paired sera of the hemagglutination inhibition reaction after vaccination)
Incidence of influenza and acute respiratory infections (ARI) | Month 1-6
  • Incidence of influenza and ARI (Month 1 - Month 6 after vaccination)
The severity and duration of registered cases of influenza and acute respiratory infections (ARI), the presence of complications | Month 1 to Month 6
  The severity and duration of registered cases of influenza and ARI, the presence of complications (Month 1 - Month 6 after vaccination)
To assess the reactogenicity of the vaccine Grippol Quadrivalent and the vaccine Grippol plus | First 7 days after vaccination
  Frequency and nature of general and local post-vaccination reactions (7-day follow-up period after vaccine administration)
Frequency and nature of SAEs | Baseline to month 6
  Frequency and nature of SAEs (Day 1-Month 6)
Frequency and nature of medically attended AEs | Baseline to month 6
  Frequency and nature of medically attended AEs (Month 1-Month 6)

CONTACTS AND LOCATIONS:
Locations (14):
- Russia (14):
  - Federal State Budgetary Research Institution "Russian research center of surgery named after academician B.V. Petrovsky", Moscow
  - State Budgetary Healthcare Institution "Children's City Clinical Hospital No.9 named after G.N. Speransky of Moscow Healthcare Department", Moscow
  - State Budgetary Health Institution of the Perm Territory "City Children's Clinical Polyclinic No. 5, Perm
  - Limited Liability Company "Clinic USI 4D", Pyatigorsk
  - Limited Liability Company Medical technology, Saint Petersburg
  - St. Petersburg State Budgetary Health Institution "Children's City Polyclinic No. 45 of the Nevsky District", Saint Petersburg
  - Limited Liability Company " Energiia Zdoroviya", Saint Petersburg
  - Limited Liability Company PiterClinica, Saint Petersburg
  - Federal State-Financed Institution Pediatric Research and Clinical Center for Infectious Diseases under the Federal Medical Biological Agency, Saint Petersburg
  - St. Petersburg State Budgetary Healthcare Institution City Polyclinic No.106 Children's Polyclinic Department No. 37, Saint Petersburg
  - State Budgetary Healthcare Institution of the Samara region "Samara Regional Children's Clinical Hospital named after N.N. Ivanova", Samara
  - Limited Liability Company Center DNK-issledovaniy, Saratov
  - Federal State Budgetary Educational Institution of Higher Education "Tyumen State Medical University" of the Ministry of Healthcare of the Russian Federation, Tyumen
  - State Autonomous Healthcare Institution of the Sverdlovsk Region "Children's City Clinical Hospital No. 11", Yekaterinburg

IPD SHARING:
Plan to Share IPD: No